CLINICAL TRIAL: NCT02046720
Title: The Influence of Age on Bispectral Index Associated With Propofol-induced Sedation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 1008181
Record Dates: First submitted 2014-01-09; First posted 2014-01-28 (Estimated); Last update posted 2016-03-23 (Estimated); Status verified 2016-03

CONDITIONS: Anesthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- propofol induced sedation (Experimental): Propofol was administered using a commercially available target-controlled infusion with an incorporated pharmacokinetic model developed by Schnider (Base Primea , Fresenius-Kabi, Brezins, FRANCE)12. The initial effect-site target concentration of propofol (0.5 μg/ml) was incremented by 0.5 μg/ml every 5 minutes to ensure equilibration between plasma concentration and effect site, until loss of eyelash reflex. From the beginning of infusion until LOER patients received no other agent besides propofol for the duration of the trial.
  Interventions: Drug: Propofol induced sedation

INTERVENTIONS:
Drug: Propofol induced sedation — Propofol was administered using a commercially available target-controlled infusion with an incorporated pharmacokinetic model developed by Schnider (Base Primea , Fresenius-Kabi, Brezins, FRANCE)12. The initial effect-site target concentration of propofol (0.5 μg/ml) was incremented by 0.5 μg/ml every 5 minutes to ensure equilibration between plasma concentration and effect site, until loss of eyelash reflex. From the beginning of infusion until LOER patients received no other agent besides propofol for the duration of the trial.
  The BIS index was compared between a young population (18 to 64 years old) and an elderly population (65 and more)
  Other Names: PIS

SUMMARY:
The bispectral index (BIS) is commonly used in anesthesia to evaluate the depth of sedation. Numerous studies in adults have shown good correlation between bispectral index values and depth of sedation regardless of the hypnotic drug used. Requirements of intravenous and inhalational hypnotic agents to suppress consciousness decrease with age. A study showed that the loss of consciousness (LOC) was obtained with lower concentrations of sevoflurane in elderly than in young adults, but at identical BIS values, so that BIS would predict depth of sedation better than drug monitoring. This result incited the use of bispectral index monitoring to overcome the significant pharmacological variability, especially in elderly. Nevertheless, another research with a comparable methodology during propofol-induced anaesthesia provided higher BIS values at LOC in elderly compared to younger patients. In these two trials, LOC was defined differently: either by absence of verbal response corresponding to loss of eyelash reflex (LOER) or by absence of response to prodding [(OAA/S) <2)]. Otherwise electromyographic activity (EMG) was not taken in account. As high EMG level (greater than 50 decibels) could create subtle artifact signal pollution without necessarily being displayed as artifacts, this would be misinterpreted by the BIS algorithm as EEG activity and assigned a spuriously increased BIS value.

The main objective of our study was to specifically evaluate BIS values according to age during propofol-induced sedation. LOC was measured by obtaining an OAA/S score <2 (OAA/S2), or a deeper sedation criterion: loss of eyelash reflex (LOER). The secondary objective was to specify the influence of EMG on the displayed BIS values and its age-related modifications.

DETAILED DESCRIPTION:
The study was approved by the ethics committee of the Saint-Etienne University Hospital. After informed consent, 70 patients over 18 years of age, ASA I to III, scheduled to undergo orthopaedic surgery under general anaesthesia were included.

Exclusion criteria were the presence of heart, respiratory, hepatic or renal failure; a psychiatric or neurological pathology, severe depression or dementia; gastro-oesophageal reflux, hiatal hernia; drug addiction or chronic alcoholism; obesity with a body mass index greater than 30.

The patients received no pre-medication. After insertion of a venous line, a Ringer's Lactate perfusion was initiated. Oxygen therapy at a rate of 4 litres per minute was administered in spontaneous ventilation. In case of hypoventilation (saturation (SaO2) <95% and/or end-tidal carbon dioxide concentration (EtCO2) >42 mmHg, manual ventilation with a mask at 10 l/min of O2 was administered.

Propofol was administered using a commercially available target-controlled infusion with an incorporated pharmacokinetic model developed by Schnider (Base Primea , Fresenius-Kabi, Brezins, FRANCE). The initial effect-site target concentration of propofol (0.5 μg/ml) was incremented by 0.5 μg/ml every 5 minutes to ensure equilibration between plasma concentration and effect site, until LOER. From the beginning of infusion until LOER patients received no other agent besides propofol for the duration of the trial.

LOC was evaluated by an independent observer using two different criteria: OAA/S score <2 (OAA/S2) corresponding to the absence of response to moderate prodding and LOER.

To minimize interactions between verbal or tactile stimulations and BIS values, BIS values were collected before evaluation of the OAA/S score and eyelash reflex check. Time to OAA/S2 and time to LOER were measured as well as corresponding brain and plasma concentrations of propofol.

Electroencephalographic activity was monitored by BIS Quatro XP platform® electrodes and a BIS VISTA™ 1.01 monitor (Aspect medical system, MA, USA). The impedance of each electrode was kept below 5 kΩ. The sensor were reapplied if the quality of the detected signal was not suitable to provide a reliable BIS score i.e a signal quality index (SQI) better than 50%. The trace was displayed in real time and calculated data (BIS, SQI, and EMG) were recorded continuously using the archiving function integrated in the monitor. A 30 second smoothing period was set to minimize the variability and sensitivity of artifacts. BIS values were validated throughout the trial by SQI values greater than 90.

Before induction and at the end of each propofol concentration level, BIS, EMG and SQI values were recorded. As soon as the OAA/S score was less than or equal to 4, the OAA/S score and eyelash reflex were evaluated every 2 minutes independently of the increase in effect-site concentration of propofol.

Arterial pressure, heart rate, SaO2, EtCO2 were measured before induction and then every 5 minutes until the end of trial. A decrease in systolic arterial pressure ≥20 was considered as hypotension, and heart rate <45 defined bradycardia.

Patients were included consecutively and assigned to one of the two groups according to their age: "young" 18 to 64 years (G1) and "elderly" aged 65 years and over (G2). As previously described, we considered that a difference of 15 units between the mean BIS values at LOC according to age was clinically pertinent.

Calculation of the required number of subjects was carried out to identify a difference of 15 units in the mean BIS value at LOC between both groups with a power of 90%, a 5% alpha risk, and an identical variability for these 2 groups (SD = 20). Thirty-five patients have to be included in each group.

The qualitative data were compared by a chi-squared test or when indicated by a Fisher's exact test. After verification of the normality of their distribution by a Kolmogorov Smirnov test, quantitative data were compared by a Student's t-test. A linear regression was used to measure the effect of age on BIS and EMG values at OAA/S2 and LOER. All the statistical analysis were performed using JMP 6 (SAS Institute Inc, Carry, NC, USA). Values p< 0.05 was considered to be statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* patients over 18 years
* ASA I to III
* scheduled to undergo orthopaedic surgery under general anaesthesia

Exclusion Criteria:

* presence of heart, respiratory, hepatic or renal failure
* psychiatric or neurological pathology
* severe depression or dementia
* gastro-oesophageal reflux
* hiatal hernia
* drug addiction or chronic alcoholism
* obesity with a body mass index greater than 30

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2010-06; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Bispectral Index (BIS) values | loss of consciousness (LOC), approximatively 20 to 30 minutes after the beginning of anesthesia
  Electroencephalographic activity was monitored by BIS Quatro XP platform® electrodes and a BIS VISTA™ 1.01 monitor (Aspect medical system, MA, USA). The impedance of each electrode was kept below 5 kΩ. The sensor were reapplied if the quality of the detected signal was not suitable to provide a reliable BIS score i.e a signal quality index (SQI) better than 50%. The trace was displayed in real time and calculated data (BIS) were recorded continuously using the archiving function integrated in the monitor. A 30 second smoothing period was set to minimize the variability and sensitivity of artifacts. BIS values were validated throughout the trial by SQI values greater than 90.

SECONDARY OUTCOMES:
the EMG component of the bispectral index value | loss of consciousness approximatively 20 to 30 minutes after the beginning of anesthesia
  Electroencephalographic activity was monitored by BIS Quatro XP platform® electrodes and a BIS VISTA™ 1.01 monitor (Aspect medical system, MA, USA). Calculated data (EMG) were recorded continuously using the archiving function integrated in the monitor. A 30 second smoothing period was set to minimize the variability and sensitivity of artifacts. The frequency of EMG will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie PASSOT, MD, Principal Investigator — CHU de Saint-Etienne
Locations (1):
- CHU de Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No